CLINICAL TRIAL: NCT04344717
Title: Pharmacokinetics of Apixaban in Patients With Short Bowel Syndrome Requiring Long Term Parenteral Nutrition
Acronym: ABSORB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: s63950
Record Dates: First submitted 2020-04-03; First posted 2020-04-14 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-11

CONDITIONS: Short Bowel Syndrome; Anticoagulation
Keywords: Apixaban; Pharmacokinetics
MeSH Terms: conditions — Short Bowel Syndrome | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Interventional, non-randomized, open label, monocentric controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Anticoagulation and teduglutide naive short bowel syndrome (Experimental): Apixaban-, vitamin K antagonist- and teduglutide naive patients with short bowel syndrome requiring long term parenteral support
  Interventions: Drug: Apixaban single dose
- Healthy volunteers (Experimental): Apixaban- and vitamin K antagonist naive healty volunteers
  Interventions: Drug: Apixaban single dose
- Short bowel syndrome on apixaban (Other): Patients with short bowel syndrome requiring long term parenteral support and taking apixaban 2.5 mg twice daily or 5 mg twice daily
  Interventions: Drug: Apixaban steady-state
- Patients with a normal gastrointestinal tract on apixaban (Other): Patients with a normal gastrointestinal tract taking apixaban 2.5 mg twice daily or 5 mg twice daily
  Interventions: Drug: Apixaban steady-state
- Anticoagulation naive short bowel syndrome on teduglutide (Experimental): Apixaban- and vitamin K antagonist naive patients with short bowel syndrome requiring long term parenteral support and initiated on teduglutide
  Interventions: Drug: Apixaban single dose

INTERVENTIONS:
Drug: Apixaban single dose — A single dose of apixaban 2.5 mg and 5 mg (wash out period of at least 7 days) will be administered and PK characteristics will be measured
  Other Names: Eliquis single dose
  Arms: Anticoagulation and teduglutide naive short bowel syndrome; Anticoagulation naive short bowel syndrome on teduglutide; Healthy volunteers
Drug: Apixaban steady-state — Steady-state apixaban PK characteristics will be measured in patients already treated with apixaban
  Other Names: Eliquis steady-state
  Arms: Patients with a normal gastrointestinal tract on apixaban; Short bowel syndrome on apixaban

SUMMARY:
Short bowel syndrome (SBS) is defined as a loss of function of the small intestine resulting in a malabsorptive disorder. In SBS, oral drug absorption may be altered due to extensive intestinal resection. It remains unclear to what extent apixaban exposure is impacted in SBS.Therefore this study tries to investigate the pharmacokinetics (PK) of apixaban in adult patients with SBS requiring long-term parenteral nutrition (PN).

ELIGIBILITY:
Inclusion criteria SBS single dose:

- patients with SBS (small bowel length of <2m after Treitz ligament) on long term (>3 months) PN or fluids who are apixaban-, vitamin K antagonist- and teduglutide naive

Inclusion criteria SBS steady-state:

- patients with SBS (small bowel length of <2m after Treitz ligament) on long term (>3 months) PN or fluids who are teduglutide naive and who are already taking apixaban 2,5 mg or 5 mg twice daily for ≥ 4 days

Inclusion criteria non-SBS single dose:

- healthy individuals without history of GI resections or other conditions associated with impaired absorption, who are apixaban- and vitamin K antagonist naive

Inclusion criteria non-SBS steady-state:

- patients without history of gastrointestinal resections or other conditions associated with impaired absorption (= controls), who are already taking apixaban 2,5 mg or 5 mg twice daily for ≥ 4 days

Exclusion criteria SBS (single dose+ steady-state):

* <18 years
* non-Dutch speaking
* recent (<6 months) major bleeds according with the International Society on Thrombosis and Haemostasis definition of major bleeding in non-surgical patients (20)
* creatinine clearance of < 15 mL/min or dialysis dependent
* liver failure classified as Child Pugh C
* total bilirubin ≥ 1.77 mg/dL (= 1,5 x upper limit of normal)
* presence of coagulopathy and a clinically relevant bleeding risk
* pregnancy or lactation
* concomitant intake of strong combined inhibitors of CYP3A4 and P-gp
* participation in a recent (<1 month) trial with an investigational product
* recent (<6 months) gastrointestinal surgery
* gastrointestinal mucosal disease interfering with absorption (e.g. radio-enteritis, inflammatory bowel disease, celiac disease, …)
* gastrointestinal fistulae
* SBS with intestinal failure resulting from gastric bypass surgery

Exclusion criteria non-SBS (single dose+ steady-state):

* <18 years
* non-Dutch speaking
* recent (<6 months) major bleeds according with the International Society on Thrombosis and Haemostasis definition of major bleeding in non-surgical patients (20)
* creatinine clearance of < 15 mL/min or dialysis dependent
* liver failure classified as Child Pugh C
* total bilirubin ≥ 1.77 mg/dL (= 1,5 x upper limit of normal)
* presence of coagulopathy and a clinically relevant bleeding risk
* pregnancy or lactation
* concomitant intake of strong combined inhibitors of CYP3A4 and P-gp
* use of prokinetics, antimotility drugs or opioids
* participation in a recent (<1 month) trial with an investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Difference in Cmax of apixaban between SBS and patients with a normal gastrointestinal tract | Through study completion, an average of 1.5 years
  To investigate the difference in peak level (Cmax) after two different single dose administrations (2,5 mg and 5 mg) of apixaban between patients with and without SBS requiring long-term PN

SECONDARY OUTCOMES:
Difference in estimated trough level (Cmin) of apixaban between SBS and patients with a normal gastrointestinal tract | Through study completion, an average of 1.5 years
  To investigate differences in estimated Cmin (12h after administration) after two different single dose administrations (2,5 mg and 5 mg) of apixaban between patients with and without SBS requiring long-term PN
Difference in time to reach Cmax (Tmax) of apixaban between SBS patients and patients with a normal gastrointestinal tract | Through study completion, an average of 1.5 years
  To investigate differences in Tmax after two different single dose administrations (2,5 mg and 5 mg) of apixaban between patients with and without SBS requiring long-term PN
Difference in exposure (AUC0-12h) of apixaban between SBS patients and patients with a normal gastrointestinal tract | Through study completion, an average of 1.5 years
  To investigate differences in AUC0-12 after two different single dose administrations (2,5 mg and 5 mg) of apixaban between patients with and without SBS requiring long-term PN
Difference in absorption rate constant of apixaban between SBS patients and patients with a normal gastrointestinal tract | Through study completion, an average of 1.5 years
  To investigate the difference in absorption rate constant between patients with and without SBS requiring long-term PN
Difference in bioavailability of apixaban between SBS patients and patients with a normal gastrointestinal tract | Through study completion, an average of 1.5 years
  To investigate the difference in bioavailability between patients with and without SBS requiring long-term PN
Difference in volume of distribution of apixaban between SBS patients and patients with a normal gastrointestinal tract | Through study completion, an average of 1.5 years
  To investigate the difference in volume of distribution between patients with and without SBS requiring long-term PN
Difference in clearance of apixaban between SBS patients and patients with a normal gastrointestinal tract | Through study completion, an average of 1.5 years
  To investigate the difference in clearance between patients with and without SBS requiring long-term PN
Difference in half-life of apixaban between SBS patients and patients with a normal gastrointestinal tract | Through study completion, an average of 1.5 years
  To investigate the difference in half-life between patients with and without SBS requiring long-term PN
To set up an optimized dosing scheme of apixaban for SBS patients | Through study completion, an average of 1.5 years
  To set up an optimized dosing scheme of apixaban, using PK modeling, for SBS patients taking into account identified covariates (eg. sex, age, race...) and PK measurements from outcome 1-9.
Difference in Cmax between SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in Cmax between SBS patients with and without teduglutide
Difference in Cmin between SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in Cmin between SBS patients with and without teduglutide
Difference in Tmax between SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in Tmax between SBS patients with and without teduglutide
Difference in AUC SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in Cmax, Cmin, Tmax, AUC, absorption rate constant, bioavailability, volume of distribution, clearance and half-life between SBS patients with and without teduglutide
Difference in AUC between SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in Cmax, Cmin, Tmax, AUC, absorption rate constant, bioavailability, volume of distribution, clearance and half-life between SBS patients with and without teduglutide
Difference in absorption rate constant between SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in absorption rate constant between SBS patients with and without teduglutide
Difference in bioavailability between SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in bioavailability between SBS patients with and without teduglutide
Difference in volume of distribution between SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in volume of distribution between SBS patients with and without teduglutide
Difference in clearance between SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in clearance between SBS patients with and without teduglutide
Difference in half-life between SBS patients with and without teduglutide | Through study completion, an average of 1.5 years
  To investigate the difference in half-life between SBS patients with and without teduglutide

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be coded according to General Data Protection Regulation

REFERENCES:
- [Background] Jeppesen PB. Spectrum of short bowel syndrome in adults: intestinal insufficiency to intestinal failure. JPEN J Parenter Enteral Nutr. 2014 May;38(1 Suppl):8S-13S. doi: 10.1177/0148607114520994. Epub 2014 Jan 31. PMID 24486858
- [Background] Santamaria MM, Villafranca JJA, Abiles J, Lopez AF, Rodas LV, Goitia BT, Navarro PU. Systematic review of drug bioavailability following gastrointestinal surgery. Eur J Clin Pharmacol. 2018 Dec;74(12):1531-1545. doi: 10.1007/s00228-018-2539-9. Epub 2018 Aug 22. PMID 30136101
- [Background] Eikelboom JW, Quinlan DJ, Hirsh J, Connolly SJ, Weitz JI. Laboratory Monitoring of Non-Vitamin K Antagonist Oral Anticoagulant Use in Patients With Atrial Fibrillation: A Review. JAMA Cardiol. 2017 May 1;2(5):566-574. doi: 10.1001/jamacardio.2017.0364. PMID 28355459